CLINICAL TRIAL: NCT06385080
Title: A Phase 1b/2, Open-label Study of Amivantamab Monotherapy and Amivantamab in Addition to Other Therapeutic Agents in Participants With Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of Amivantamab Alone or in Addition to Other Treatment Agents in Participants With Head and Neck Cancer
Acronym: OrigAMI-4
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61186372HNC2002; 61186372HNC2002 (Other: Janssen Research & Development, LLC); 2023-508418-40-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-04-23; First posted 2024-04-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — amivantamab; pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: Amivantamab Monotherapy (Dose Expansion) (Experimental): Participants will receive subcutaneous injection of amivantamab monotherapy 1600 milligrams (mg) (2240 mg, if body weight >=80 kilograms [kg]) on Cycle 1 Day 1 and 2400 mg (3360 mg, if body weight >=80 kg) once every week (q1w) for the remainder of Cycle 1 (Days 8 and 15), and every 3 weeks (q3w) from Cycle 2 onwards.
  Interventions: Biological: Amivantamab
- Cohort 2: Amivantamab + Pembrolizumab (Dose Expansion Including Safety Run-in) (Experimental): Participants will receive subcutaneous injection of amivantamab 1600 mg (2240 mg, if body weight >=80 kg) on Cycle 1 Day 1 and 2400 mg (3360 mg, if body weight >=80 kg) q1w for the remainder of Cycle 1 (Days 8 and 15), and q3w from Cycle 2 onwards, along with intravenous (IV) injection of pembrolizumab 200 mg q3w (on Day 1 of each 21-day cycle).
  Interventions: Biological: Amivantamab; Biological: Pembrolizumab
- Cohort 3A (Dose Confirmation): Amivantamab + Paclitaxel (Experimental): Participants will receive subcutaneous injection of amivantamab 1600 mg (2240 mg, if body weight >=80 kg) on Cycle 1 Day 1 and 2400 mg (3360 mg, if body weight >=80 kg) q1w for the remainder of Cycle 1 (Days 8 and 15), and q3w from Cycle 2 onwards, along with intravenous injection of paclitaxel 175 mg/m^2 q3w (on Day 1 of each 21-day cycle) in dose confirmation Cohort 3A. The recommended Phase 2 combination dose (RP2CD) of amivantamab will be determined in conjunction with study evaluation team (SET) in this dose confirmation Cohort 3A.
  Interventions: Biological: Amivantamab; Drug: Paclitaxel
- Cohort 3B (Dose Expansion): Amivantamab + Paclitaxel (Experimental): Participants will receive subcutaneous injection of amivantamab at the determined RP2CD in addition to intravenous injection of paclitaxel 175 mg/m^2 q3w (on Day 1 of each 21-day cycle) as confirmed by SET in Cohort 3A.
  Interventions: Biological: Amivantamab; Drug: Paclitaxel
- Cohort 4: Amivantamab Monotherapy (Experimental): Participants will receive subcutaneous injection of amivantamab monotherapy 1600 mg (2240 mg, if body weight >=80 kg) on Cycle 1 Day 1 and 2400 mg (3360 mg, if body weight >=80 kg) q1w for the remainder of Cycle 1 (Days 8 and 15), and q3w from Cycle 2 onwards.
  Interventions: Biological: Amivantamab
- Cohort 5: Pembrolizumab + Amivantamab + Carboplatin (Dose Expansion) (Experimental): Participants will receive subcutaneous injection of amivantamab 1600 mg (2240 mg, if body weight >=80 kg) on Cycle 1 Day 1 and 2400 mg (3360 mg, if body weight >=80 kg) q1w for the remainder of Cycle 1 (Days 8 and 15), and q3w from Cycle 2 onwards in addition to intravenous injection of pembrolizumab 200 mg on Day 1 of each cycle, and carboplatin (area under the concentration-time curve [AUC] 5 milligram per milliliter [mg/ml]*min) q3w on Day 1 of Cycles 1-6.
  Interventions: Biological: Amivantamab; Biological: Pembrolizumab; Drug: Carboplatin
- Cohort 6: Amivantamab + Pembrolizumab (Experimental): Participants will receive subcutaneous injection of amivantamab 1600 mg (2240 mg, if body weight >=80 kg) on Cycle 1 Day 1 and 2400 mg (3360 mg, if body weight >=80 kg) q1w for the remainder of Cycle 1 (Days 8 and 15), and q3w from Cycle 2, along with intravenous injection of pembrolizumab 200 mg q3w (on Day 1 of each 21-day cycle) (Neoadjuvant Phase). In the adjuvant phase, pembrolizumab IV (200 mg) will be administered q3w from Adjuvant Cycle 1 Day 1 to Adjuvant Cycle 15 Day 1 and amivantamab SC 2,400 mg (3,360 mg for >80 kg) will be administered q3w from Adjuvant Cycle 4 Day 1 to Adjuvant Cycle 15 Day 1.
  Interventions: Biological: Amivantamab; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Amivantamab — Amivantamab will be administered subcutaneously.
  Other Names: JNJ-61186372
Biological: Pembrolizumab — Pembrolizumab will be administered intravenously.
  Other Names: KEYTRUDA
  Arms: Cohort 2: Amivantamab + Pembrolizumab (Dose Expansion Including Safety Run-in); Cohort 5: Pembrolizumab + Amivantamab + Carboplatin (Dose Expansion); Cohort 6: Amivantamab + Pembrolizumab
Drug: Paclitaxel — Paclitaxel will be administered intravenously.
  Other Names: TAXOL
  Arms: Cohort 3A (Dose Confirmation): Amivantamab + Paclitaxel; Cohort 3B (Dose Expansion): Amivantamab + Paclitaxel
Drug: Carboplatin — Carboplatin will be administered intravenously.
  Other Names: PARAPLATIN
  Arms: Cohort 5: Pembrolizumab + Amivantamab + Carboplatin (Dose Expansion)

SUMMARY:
The purpose of this study is to determine safety and preliminary efficacy of amivantamab monotherapy, amivantamab in addition to pembrolizumab, amivantamab in addition to paclitaxel and amivantamab in addition to pembrolizumab and carboplatin in participants with recurrent/metastatic head and neck cancer. The study will also confirm the recommended Phase 2 combination dose (RP2CD) for amivantamab in addition to paclitaxel. The safety and preliminary efficacy of amivantamab in addition to pembrolizumab will also be determined in perioperative (before and after surgery) setting in participants with resectable locally advanced head and neck squamous cell carcinoma (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Cohorts 1 to 5: Have histologically or cytologically confirmed recurrent/metastatic head and neck squamous cell carcinoma (R/M HNSCC) that is considered incurable by local therapies or for Cohort 6: have histologically or cytologically confirmed locally advanced (L/A) HNSCC that is considered curable by surgery Acceptable prior lines of therapy will be determined according to specific cohort 1, 2, 3A and 3B: (a) The eligible primary tumor locations are the oropharynx, oral cavity, hypopharynx, or larynx; (b) Any known p16 status of tumor must be negative (Note: All participants with an oropharyngeal tumor must have results of p16 status, per local testing); (c) Participants must provide local testing results of programmed cell death ligand 1 (PD-L1) status, if available; Cohort 4: (d) Patients must have primary tumor location in oropharynx. Unknown primary tumors are not included (e) Primary tumor must be HPV-positive, confirmed by positive p16 test or high-risk human papillomavirus (HPV) in-situ hybridization (ISH) in tissue (current or archival) (f) Participants must provide local testing results of PD-L1 status, if available; Cohort 5 (g) The eligible primary tumor locations are the oropharynx, oral cavity, hypopharynx, or larynx; (h) HPV status must be known (either positive or negative) for patients with primary tumor location in oropharynx with p16 test or high-risk HPV ISH in tissue; (i) Participants must provide local testing results of PD-L1 status; Cohort 6: (j) The eligible primary tumor locations are the oropharynx, oral cavity, hypopharynx, or larynx; (k) Any known p16 status of tumor must be negative Note: All participants with an oropharyngeal tumor must have results of p16 status, per local testing Participants must provide local testing results of PD-L1 status (l) Participants must have Stage III or IVa disease (American Joint Committee on Cancer Staging Manual, 8th edition). Participants must have resectable disease
* Participants in Cohorts 1, 2, 3B, 4 and 5 must have measurable disease according to RECIST version 1.1. Participants in Cohort 3A and Cohort 6 must have evaluable disease (defined as having at least 1 non-target lesion according to RECIST version 1.1.
* Cohorts 1, 2, 3A, 3B, 4, and 5 only: Toxicities from previous anticancer therapies should have resolved to baseline levels or to Grade 1 or less prior to the first dose of study treatment (except for alopecia or post-radiation skin changes [any grade], Grade less than or equal to [<=]2 peripheral neuropathy and Grade <=2 hypothyroidism stable on hormone replacement)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Participant must have adequate organ and bone marrow function as follows, without history of red blood cell transfusion, platelet transfusion, or use of granulocyte colony-stimulating factor within 7 days prior to the date of the laboratory test.

Participants should have: a) Hemoglobin >=9 grams per deciliter (g/dL); b) Neutrophils >=1.5 x 10^3/mcg; c) Platelets >=100 x 10^3/mcg

Exclusion Criteria:

* Uncontrolled illness including any medical history or current (non-infectious) interstitial lung disease (ILD)/ pneumonitis/ pulmonary fibrosis, or where suspected ILD/pneumonitis/pulmonary fibrosis cannot be ruled out by imaging at screening
* Participant with untreated brain metastases leptomeningeal disease, or spinal cord compression not definitively treated with surgery or radiation
* Participant with a history of clinically significant cardiovascular disease
* Received prior chemotherapy, targeted cancer therapy, immunotherapy, or treatment with an investigational anticancer agent within 2 weeks or 4 half-lives, whichever is longer, before the first administration of study treatment. The maximum required washout is 28 days
* Received radiotherapy for palliative purposes within 7 days of the first administration of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-12-27 (Estimated); Study Completion 2032-12-27 (Estimated)

PRIMARY OUTCOMES:
Cohorts 1, 2, 3B, 4 and 5: Objective Response Rate | 2 years and 2 months
  ORR is defined as the proportion of participants who achieve either a partial response (PR) or complete response (CR), as defined by investigator assessment using Response Criteria in Solid Tumors (RECIST) version 1.1.
Cohort 3A: Number of Participants With Dose-limiting Toxicities (DLT) | Up to 21 days
  Number of participants with DLTs will be reported. A DLT is defined as any of the following: treatment delay of greater than (>) 28 days due to unresolved toxicity, non-hematologic toxicity of Grade 3 or higher, hematologic toxicity of Grade 4 neutropenia persisting for >7 days or Grade 3 or higher thrombocytopenia with clinically significant bleeding or neutropenic fever of any grade, and liver enzyme elevation.
Cohort 3A: Number of Participants With Treatment-emergent Adverse Events (TEAEs) as a Measure of Severity | 2 years and 1 month
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment. Severity of TEAEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (mild) to Grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening, and Grade 5= death related to adverse event.
Cohort 6: Major Pathologic Response (MPR) | 2 years and 2 months
  The participants who achieve MPR at the time of surgery.

SECONDARY OUTCOMES:
Cohorts 1, 2, 3B, 4 and 5: Duration of Response (DoR) | 2 years and 2 months
  DoR is defined as the time from the date of first documented response (PR or CR) until the date of documented progression or death, whichever comes first, for participants who have PR or CR.
Cohorts 1, 2, 3B, 4 and 5: Clinical Benefit Rate (CBR) | 2 years and 2 months
  CBR is defined as the percentage of participants achieving a confirmed complete or partial response, or durable stable disease (the second disease assessment) as defined by RECIST version 1.1.
Cohorts 1, 2, 3B, 4 and 5: Progression-free Survival (PFS) | 2 years and 2 months
  PFS is defined as the time from the first administration of study treatment until the date of objective disease progression or death, whichever comes first, based on investigator assessment using RECIST version 1.1.
Cohorts 1, 2, 3B, 4, 5 and 6: Overall Survival (OS) | 2 years and 2 months
  OS is defined as the time from the first administration of study treatment until the date of death due to any cause.
Cohorts 1, 2, 3B, 4, 5 and 6: Number of Participants With Treatment-emergent Adverse Events (TEAEs) as a Measure of Severity | 2 years and 1 month
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment. Severity of TEAEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse events.
Cohort 1 and 4: Maximum Observed Serum Concentration (Cmax) of Amivantamab | Predose up to 168 hours post dose on Day 1
  Cmax is defined as maximum observed serum concentration of amivantamab.
Cohort 1 and 4: Time to Maximum Observed Serum Concentration (Tmax) of Amivantamab | Predose up to 168 hours post dose on Day 1
  Tmax is defined as time to maximum observed serum concentration of amivantamab.
Cohort 1 and 4: Area Under the Serum Concentration Curve Verses Time Curve From Time t1 to t2 (AUC[t1-t2]) of Amivantamab | Predose up to 168 hours post dose on Day 1
  AUC(t1-t2) is defined as area under the serum concentration versus time curve from time t1 to time t2 of amivantamab.
Cohort 1 and 4: Area Under the Curve From Time Zero to tau (AUC[0-tau]) of Amivantamab | Predose up to 168 hours post dose on Day 1
  AUC(0-tau) is defined as area under the curve from time 0 to tau hours of amivantamab.
Cohort 1 and 4: Trough Serum Concentration (Ctrough) of Amivantamab | Predose up to 168 hours post dose on Day 1
  Ctrough is defined as the serum concentration of amivantamab.
Cohort 1 and 4: Accumulation Ratio (R) of Amivantamab | Predose up to 168 hours post dose on Day 1
  Accumulation ratio (R) is calculated as area under the serum concentration-time curve from time zero to 168 hours (AUC[0-168]) value at Cycle 2 Day 1 dose divided by AUC(0-168) value after Cycle 1 Day 1 amivantamab dose.
Cohort 6: Event-Free Survival (EFS) | 2 years and 2 months
  EFS is defined as the time from the first administration of study treatment until the date of radiographic disease progression, local or distant progression or recurrence as assessed with imaging or biopsy as indicated, or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (55):
- United States (14):
  - University of California at San Diego Moores Cancer Center, La Jolla, California
  - University of Colorado Denver Anschultz Medical Campus, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
- China (6):
  - Beijing Cancer Hospital of Peking University, Beijing
  - West China School of Medicine/West China Hospital, Sichuan University, Cheng Du Shi
  - Linyi Cancer Hospital, Linyi
  - Fudan Cancer Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
- France (5):
  - Institut Sainte Catherine, Avignon
  - Centre Oscar Lambret, Lille
  - CHU Nantes, Nantes
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Landeshauptstadt Stuttgart, Stuttgart
- Japan (2):
  - Aichi Cancer Center, Nagoya
  - Tokyo Medical University Hospital, Tokyo
- Malaysia (2):
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Onkologii Instytut im M Sklodowskiej Curie Oddzial w Gliwicach, Gliwice
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hosp Univ Vall D Hebron, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (7):
  - Addenbrooke's Hospital, Cambridge
  - The Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - Royal Marsden Hospital, London
  - Imperial College London and Imperial College Healthcare NHS Trust, London
  - University College London Hospitals, London
  - The Christie Nhs Foundation Trust, Manchester
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency